CLINICAL TRIAL: NCT03501251
Title: Efficacy and Safety of Ascending Dosages of Moxidectin and Moxidectin-albendazole Against Trichuris Trichiura in Adolescents: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Ascending Dosages of Moxidectin and Moxidectin-albendazole Against Trichuris Trichiura
Acronym: MOXIDOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Principal Investigator, Jennifer Keiser, Principal Investigator, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOXI_DOSE_PEMBA
Record Dates: First submitted 2018-03-01; First posted 2018-04-18 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Trichuris Trichiura; Infection
MeSH Terms: conditions — Trichuriasis | interventions — moxidectin; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will receive placebos. Outcome assessors and caregivers will not have access to the list of children allocated to each treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Moxidectin 8 mg (Experimental): A single tablet of 8 mg of moxidectin
  Interventions: Drug: Moxidectin 8mg
- Moxidectin 8 mg + Albendazole (Experimental): A single tablet of 8 mg of moxidectin plus a single tablet of albendazole (400 mg)
  Interventions: Drug: Moxidectin 8 mg + albendazole 400 mg
- Moxidectin 16 mg (Experimental): Two tablets of 8 mg of moxidectin ( = 16 mg)
  Interventions: Drug: Moxidectin 16 mg
- Moxidectin 16 mg + Albendazole (Experimental): Two tablets of 8 mg of moxidectin ( = 16 mg) plus a single tablet of albendazole (400 mg)
  Interventions: Drug: Moxidectin 16 mg + albendazole 400 mg
- Moxidectin 24 mg (Experimental): Three tablets of 8 mg of moxidectin ( = 24 mg)
  Interventions: Drug: Moxidectin 24 mg
- Moxidectin 24 mg + Albendazole (Experimental): Three tablets of 8 mg of moxidectin ( = 24 mg) plus a single tablet of albendazole (400 mg)
  Interventions: Drug: Moxidectin 24 mg + albendazole 400 mg
- Placebo (Placebo Comparator): A single tablet of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Moxidectin 8mg — Participants will receive the tablet with clean water and a package of biscuits.
  Arms: Moxidectin 8 mg
Drug: Moxidectin 8 mg + albendazole 400 mg — Participants will receive the tablets with clean water and a package of biscuits.
  Arms: Moxidectin 8 mg + Albendazole
Drug: Moxidectin 16 mg — Participants will receive the tablets with clean water and a package of biscuits.
  Arms: Moxidectin 16 mg
Drug: Moxidectin 16 mg + albendazole 400 mg — Participants will receive the tablets with clean water and a package of biscuits.
  Arms: Moxidectin 16 mg + Albendazole
Drug: Moxidectin 24 mg — Participants will receive the tablets with clean water and a package of biscuits.
  Arms: Moxidectin 24 mg
Drug: Moxidectin 24 mg + albendazole 400 mg — Participants will receive the tablets with clean water and a package of biscuits.
  Arms: Moxidectin 24 mg + Albendazole
Other: Placebo — Participants will receive the tablet with clean water and a package of biscuits.
  Arms: Placebo

SUMMARY:
The study rationale is to provide evidence on effective doses of moxidectin and/or moxidectin-albendazole in adolescents (16-18 years old) infected with Trichuris trichiura. The study will take place on Pemba Island, Tanzania.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 16 to 18 years, inclusive
2. Written informed consent/assent signed from parent/guardian
3. Positive for T. trichiura by at least two slides of the quadruple Kato-Katz thick smears and infection intensities of at least 100 eggs per gram of stool (EPG)
4. Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and approximately three weeks after treatment (follow-up).

Exclusion Criteria:

1. Presence of acute or uncontrolled systemic illnesses (e.g. severe anemia, infection, clinical malaria) as assessed by a medical doctor, upon initial clinical assessment.
2. Known or reported history of chronic illness such as HIV, acute or chronic hepatitis, cancer, diabetes, chronic heart disease or renal disease.
3. Prior treatment with anthelmintics (eg, diethylcarbamazine [DEC], suramin, ivermectin or albendazole) within 4 weeks before planned test article administration.
4. Received any investigational drugs or investigational devices within 4 weeks before administration of test article that may confound safety and/or efficacy assessments.
5. Known or suspected allergy to moxidectin, ivermectin or albendazole or other compounds related to these classes of medication.
6. Pregnant (urine testing) or breastfeeding women

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Cure rate against Trichuris trichiura | 6 weeks
  Conversion from being Trichuris trichiura-egg positive pre-treatment to egg negative post-treatment. Since this might be influenced by infection intensity, treatment groups will be equally balanced in terms of infection intensity by 2 levels of baseline infection intensity (light infections and moderate/heavy infections).

SECONDARY OUTCOMES:
Egg Reduction Rate of the different drug regimens against Trichuris trichiura | 6 weeks
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Cure rate of the different drug regimens against Ascaris lumbricoides | 6 weeks
  Conversion from being Ascaris lumbricoides-egg positive pre-treatment to egg negative post-treatment.
Egg Reduction Rate of Ascaris lumbricoides | 6 weeks
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Cure rate against hookworm | 6 weeks
  Conversion from being hookworm-egg positive pre-treatment to egg negative post-treatment.
Egg Reduction Rate of hookworm | 6 weeks
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Number of adverse events at 5 time points | 6 weeks
  Patients will be kept for observation for at least 3 hours following treatment for any acute adverse events. During the reporting period, any unfavorable changes in the subject's condition will be recorded as adverse events, whether reported by the subject or observed by the Investigator. In case of any abnormal finding, the local study physician will perform a full clinical examination and findings will be recorded. An emergency kit will be available on site to treat any medical conditions that warrant urgent medical intervention. In addition, patients will be also interviewed by a nurse and/or a physician about the occurrence of adverse events 24, 48 and 72 hours post-treatment using a questionnaire. Finally, upon collection of the first follow-up stool sample participants will be re-questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory Ivo de Carneri, P.O. Box 122, Chake Chake, Pemba, Tanzania

REFERENCES:
- [Derived] Keller L, Palmeirim MS, Ame SM, Ali SM, Puchkov M, Huwyler J, Hattendorf J, Keiser J. Efficacy and Safety of Ascending Dosages of Moxidectin and Moxidectin-albendazole Against Trichuris trichiura in Adolescents: A Randomized Controlled Trial. Clin Infect Dis. 2020 Mar 3;70(6):1193-1201. doi: 10.1093/cid/ciz326. PMID 31044235